CLINICAL TRIAL: NCT03686657
Title: A 26-week Single Site, Randomized, Double-blind, Active-controlled, Parallel Group, Human PoC Study to Evaluate Superiority of RK-01, Valsartan Plus Celecoxib Addon to Metformin Versus Metformin Alone in Type 2 Diabetes Patients
Brief Title: Evaluation of Superiority of Valsartan+Celecoxib+Metformin Over Metformin Alone in Type 2 Diabetes Patients
Acronym: RESILIENCE
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ARKAY Therapeutics (Industry)
Collaborators: Albany Medical College (Other); Myopharm Limited (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TriGlytza (RK-01) Prototype
Record Dates: First submitted 2018-09-23; First posted 2018-09-27 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Type 2 Diabetes; High Blood Pressure; Arthritis; Obesity
Keywords: Diabetes; Obesity; FPG; Beta cell function index; HbA1c; Atherogenic index
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension; Arthritis; Obesity; Diabetes Mellitus | interventions — Metformin; Valine; Carboxylesterase; Valsartan; Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Healthy adults with NGT (No Intervention): Healthy adults with normal glucose tolerance (NGT) and beta cell function will be administered placebo.
- Metformin-Drug naive patients & Patients with inadequate glycemic control with Metformin (Active Comparator): Patients receive metformin once daily
  Interventions: Drug: Metformin
- RK-01 Low (Experimental): Patients receive valsartan, celecoxib and metformin (low dose) once daily
  Interventions: Drug: Val, Cel and Met XR Low
- RK-01 High (Experimental): Patients receive valsartan, celecoxib and metformin (high dose) once daily
  Interventions: Drug: Val, Cel and Met XR High

INTERVENTIONS:
Drug: Metformin — 1000 mg metformin-HCL XR once-a-day or maintenance dose of metformin for 26 weeks
  Other Names: Glucophage; Glucophage XR
  Arms: Metformin-Drug naive patients & Patients with inadequate glycemic control with Metformin
Drug: Val, Cel and Met XR Low — 500 mg metformin-HCL XR plus 100 mg celecoxib once-a-day in the morning and 160 mg valsartan 6 hours later once-a-day in the afternoon for 26 weeks.
  Other Names: Diovan; Celebrex; Glucophage XR; RK-01
  Arms: RK-01 Low
Drug: Val, Cel and Met XR High — 1000 mg metformin-HCL XR plus 200 mg celecoxib once-a-day in the morning and 320 mg valsartan once-a-day 6 hours later in the afternoon for 26 weeks.
  Other Names: Diovan; Celebrex; Glucophage XR; RK-01
  Arms: RK-01 High

SUMMARY:
Evaluation of safety, tolerability and superiority of RK-01, a valsartan plus celecoxib dual add-on to metformin-HCL XR over metformin in newly diagnosed and obese adult type 2 diabetes patients with high blood pressure, arthritis and inadequate glycemic control with metformin monotherapy, diet and exercise over 26 weeks of treatment.

Objective: To assess effect of RK-01 on HbA1c levels, beta cell function and insulin resistance with co-administration of valsartan, celecoxib and metformin-HCl XR relative to metformin monotherapy.

Hypothesis: After 26 weeks of treatment with valsartan, celecoxib and metformin-HCl XR provides greater improvements in glycemic, inflammatory and atherogenic parameters compared to metformin monotherapy.

DETAILED DESCRIPTION:
PRIMARY:

In patients with type 2 diabetes with inadequate glycemic control with metformin monotherapy:

Objective: To assess effect of RK-01 on HbA1c levels, beta cell function and insulin resistance with co-administration of valsartan, celecoxib and metformin-HCl XR relative to metformin monotherapy. Improvements in glycemic, inflammatory and atherogenic parameters including beta cell function relative to adult healthy volunteers with normal glucose tolerance (NGT) treated with placebo for 26 weeks will also be assessed. An interim study assessment will also be performed after 12 weeks of treatment.

Hypothesis: After 26 weeks of treatment with valsartan, celecoxib and metformin-HCl XR provides greater improvements in glycemic, inflammatory and atherogenic parameters compared to metformin monotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, Age: >18 to 70 years at the time of screening visit.
2. Women of childbearing potential (WOCBP) must have negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent of HCG) within 24 hours prior to the start of the study.
3. Women must not be breastfeeding.
4. HbA1c≥8.0
5. Patients with inadequate blood glucose control with Metformin defined as a central laboratory glycosylated hemoglobin (HbA1c) >8.0 and <10.5 obtained at the screening visit. Metformin-HCl monotherapy was inadequate 3 months prior to the study as indicated by the lack of decrease and/or an increase in the A1c level.

   Newly diagnosed drug naïve patients as defined by HbA1c>7.0 at the screening visit. Drug naïve subjects diagnosed with type 2 diabetes within 6 months of diagnosis will be considered and selected.

   About half the patients are expected to be newly diagnosed in the study.
6. Drug naive as well as osteoarthritis patients with Type 2 diabetes receiving a non-aspirin pain reliever (e.g. acetaminophen) or an NSAID (e.g. Naproxen).
7. Max/maintenance dose Metformin. Subjects should have been taking the same daily dose of metformin for at least 8 weeks prior to the enrollment visit and subjects not receive these other antihyperglycemic medications within the 12 weeks prior to screening (except for short-term use of insulin [≤7 days] during concomitant illness or other stress).
8. Patients with >25% AIRg at 2 minutes and 10 minutes.
9. RAS blocker naïve patients
10. 2-Hour OGTT ≥200 mg/dL
11. FPG ≥140 mg/dL
12. BMI ≥30
13. Impaired first phase and second phase of insulin secretion
14. BP ≥140/90 mm Hg (These patients might be on an anti-hypertensive drug)
15. Non-fasting laboratory glucose >200 mg/dL with symptoms of polydipsia, polyuria and/or Polyphagia
16. eGFR ≥ 60 ml/min/1.73m2

Exclusion Criteria:

1. Age >70
2. Patients with Type 1 diabetes, Screen for GAD (Glutamic acid decarboxylase) antibodies at the time of screening visit. To rule out latent autoimmune diabetes in adults (LADA), screening for other diabetes-related antibodies, such as insulinoma-associated protein (IA-2 and IA-2 beta), zinc transporter-8 (ZnT8), islet cell antibodies (ICA) or insulin autoantibody (IAA) will also be considered.
3. Pregnant women
4. Patients with a history of Ketoacidosis.
5. Subjects at serious risk of gastrointestinal (GI) adverse events (e.g. current or recent history of GI bleeding ulceration, or perforation).
6. Subjects with a planned radiologic study with intravenous contrast, surgery, or other planned procedures that may predispose them to metformin-associated lactic acidosis.
7. Insulin dependent: <25% Beta-cell function: AIRg (Acute insulin response to glucose after 2 min and 10 min after glucose injection) INSULIN DEPENDENT STATE.
8. Patients with a history of uncontrolled hyperglycemia >15.0 mmol/L (280 mg/dL) after an overnight fast that required rescue therapy.
9. Patients with uncontrolled hyperglycemia >15.0 mmol/L (280 mg/dL) after an overnight fast that required rescue therapy during week 1-3 Metformin-HCl monotherapy or RK-01 therapy.
10. eGFR, impaired kidney function < 60 ml/min/1.73m2.
11. Poor metabolizers of Cyp450 2C9 to avoid very high concentration (Since Cytochrome 450 2C9 is responsible for the metabolism of both Valsartan and Celecoxib, patients who are known or suspected to be poor Cyp450 2C9 metabolizers based on previous history will be excluded from the study).
12. Any of the following cardiovascular (CV)/Vascular diseases within 3 months of the enrollment visit:

    1. Myocardial infarction (MI)
    2. Cardiac surgery or revascularization (coronary artery bypass surgery, Coronary Artery Bypass Graft [(CABG]/Percutaneous transluminal coronary angioplasty (PTCA)].
    3. Unstable angina
    4. Unstable congestive heart failure (CHF)
    5. Transient ischemic attack (TIA) or significant cerebrovascular disease
    6. Unstable or previously diagnosed arrhythmia
    7. Congestive heart failure, defined as New York Heart Association (NYHA) Class III and IV, unstable or acute heart failure and/or known left ventricular ejection fraction of ≤40%.
    8. Acute coronary syndrome, stroke or transient ischemic attack within 3 months prior to the informed consent.
13. Previous bariatric surgery
14. Treatment with anti-obesity drugs within 3 months prior to consent
15. Patients with COPD
16. Patients with liver disease
17. Patients with renal disease
18. Patients with autoimmune diseases e.g. Lupus, Psoriasis
19. Patients with HIV/AIDS
20. Patients with diabetes-related complications
21. Patients with Hematological and Oncological Diseases/Conditions
22. Hemoglobin <11.0 g/dL (110 g/L) for men; hemoglobin <10.0 g/dL (100 g/L) for women
23. Patients with chronic disease e.g. Cancer, Epilepsy, Alzheimer, Parkinson, Asthma
24. Abnormal free T4
25. Patients with serious infection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2025-10-10 (Estimated); Primary Completion 2028-11-26 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in glycosylated Hemoglobin (HbA1c) for metformin background patients | Baseline and 26 weeks
  Glycosylated hemoglobin (HbA1c) is a measurement of the percentage of hemoglobin that is glycated. The change from baseline is calculated as the week 26 HbA1c minus the baseline HbA1c. Since HbA1c is measured as a percentage, the change from baseline is also a percentage.
Change in glycosylated Hemoglobin (HbA1c) for treatment naive patients | Baseline and 26 weeks
  Glycosylated hemoglobin (HbA1c) is a measurement of the percentage of hemoglobin that is glycated. The change from baseline is calculated as the week 26 HbA1c minus the baseline HbA1c. Since HbA1c is measured as a percentage, the change from baseline is also a percentage.
Change from baseline in acute insulin response to glucose (AIRg) for metformin background patients | Baseline and 26 weeks
  Change in baseline in acute insulin response to glucose at week 26
Change from baseline in acute insulin response to glucose (AIRg) for treatment naive patients | Baseline and 26 weeks
  Change in baseline in acute insulin response to glucose at week 26

SECONDARY OUTCOMES:
Change in glycosylated Hemoglobin (HbA1c) to <7.0% | Baseline and 26 weeks
  Glycosylated hemoglobin (HbA1c) is a measurement of the percentage of hemoglobin that is glycated. The change from baseline is calculated as the week 26 HbA1c minus the baseline HbA1c. Since HbA1c is measured as a percentage, the change from baseline is also a percentage. Percentage of subjects achieving a therapeutic glycemic response, defined as HbA1c <7.0%.
Change from baseline in Body weight | Baseline and 26 weeks
  Change in body weight at week 26
Change from baseline in fasting plasma glucose | Baseline and 26 weeks
  Change in baseline in fasting plasma glucose at week 26
Change from baseline in Beta-cell function Index | Baseline and 26 weeks
  Change in baseline in beta cell function index at week 26. Beta-cell function Index is a measure of their capacity to respond to elevated blood glucose levels
Change from baseline in insulin sensitivity index (ISI or Si) | Baseline and 26 weeks
  Change in baseline in insulin sensitivity at week 26
Change from baseline in glycosylated albumin (GA): glycosylated Hemoglobin A1c (HbA1c) ratio | Baseline and 26 weeks
  Change in baseline in glycosylated albumin (GA): glycosylated Hemoglobin A1c (HbA1c) at week 26. GA:HbA1c ratio provides a measure of post-prandial excursion
Change from baseline in HOMA2-b% | Baseline and 26 weeks
  Change in baseline in HOMA of Beta-cell function index at week 26
Change from baseline in HOMA-IR | Baseline and 26 weeks
  Change in baseline in HOMA-IR at week 26. HOMA-IR is a measure of insulin resistance.
Leptin/Adiponectin ratio | Baseline and 26 weeks
  Change in baseline in Leptin/Adiponectin ratio. Indicator of insulin resistance
Change from baseline in Atherogenic Index (AI) | Baseline and 26 weeks
  Change in baseline in Atherogenic Index at week 26. Atherogenic Index (AI) is a predictor of cardiovascular risk
Change from baseline in glycosylated albumin (GA) | Baseline and 26 weeks
  Change in baseline in glycosylated albumin (GA) at week 26
Change from baseline in Leptin | Baseline and 26 weeks
  Change in baseline in Leptin at week 26
Change from baseline in Adiponectin | Baseline and 26 weeks
  Change in baseline in Adiponectin at week 26

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Kumar, Ph.D., Study Director — ARKAY Therapeutics
Locations (1):
- Albany Medical College, Albany, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
Study results will be published on clinicaltrials.gov as well as a medical journal. We also plan to present the results at a conference such as American Diabetes Association's Scientific Sessions.